CLINICAL TRIAL: NCT05081973
Title: A Model for Predicting Extubation Success Based on the "Extubation Readiness Estimator" and Lung Ultrasonography Score in Premature Babies
Brief Title: A Model for Predicting Extubation Success in Premature Babies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Collaborators: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: MarmaraU_Neonatal
Record Dates: First submitted 2021-09-23; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Neonatal Respiratory Failure; Invasive Mechanical Ventilation; Extubation Failure
Keywords: Neonate; Extubation Failure; Lung Ultrasonography Score; Extubation Readiness Estimator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intubated preterm infants: Infants with a birth weight < 1250 grams who have required endotracheal tube and mechanical ventilation within the first 7 days of life, and have been on an invasive mechanical ventilator for at least 48 hours, and have not completed 60 days after birth, and have met the traditional extubation criteria of the institution, and have been considered for elective extubation for the first time.
  Interventions: Other: A model for predicting extubation success based on extubation readiness estimator and lung ultrasonography score

INTERVENTIONS:
Other: A model for predicting extubation success based on extubation readiness estimator and lung ultrasonography score — Parameters to be recorded before and after extubation to create a "new dual extubation model" from all babies who met the extubation criteria included in the study:
  1. "Lung ultrasound score": Lung ultrasound will be performed prior to the extubation and after the extubation. Lung aeration will be scored based on three chest areas for each side (upper anterior, lower anterior and lateral) and a score of 0 to 3 points will be given for each area (Total score ranges from 0 to 18 points).
  2. "Probability of Successful Extubation": It will be calculated by extubation readiness estimator provided by the website named http://extubation.net/.
  This parameter will be calculated only 1 hour prior to the scheduled extubation time.

SUMMARY:
Invasive mechanical ventilation is a life-saving treatment in critically ill newborns with respiratory failure. However, continuing this treatment for a long time may have negative consequences, especially bronchopulmonary dysplasia (BPD) secondary to mechanotrauma. For this reason, it is essential to terminate the mechanical ventilation treatment at the most appropriate time.

About half of the extremely preterm babies may fail extubation even if the clinical criteria traditionally used for extubation are met. Unsuccessful extubation is associated with increased intraventricular bleeding, death, BPD, death or BPD, longer duration of ventilator support.

When respiratory failure and lung pathologies of extremely preterm babies begin to improve, the target for mechanical ventilation should be early and successful extubation. Currently, the decision to extubate a preterm baby is primarily based on clinical judgment. Only a few studies that showed the low predictive value and limited utility using different measures have evaluated readiness for extubation. Lung ultrasonography (USG) is a noninvasive bedside technique that has been found useful for predicting the success of weaning from the ventilator in adults; however, very little data are available in neonates. In a recently published study, it was proposed an extubation readiness estimation tool based on clinical and demographic data of preterm babies who were attempted elective extubation.

The researchers' hypothesis is that the use of a model based on extubation success scoring and lung USG scoring before extubation reduces the failure of the first extubation attempt in very low birth weight infants. The aim of the study is to evaluate the value of using an integrated model based on pre-extubation "extubation readiness predictor" and lung USG scoring to predict extubation success in preterm babies undergoing invasive mechanical ventilation.

DETAILED DESCRIPTION:
Long-term invasive mechanical ventilation may have detrimental effects in preterm infants, although it is a life-saving treatment in critically ill newborns with respiratory failure. (e.g. bronchopulmonary dysplasia (BPD), superimposed bacterial infections and colonization, air leak, etc.). For this reason, it is essential to terminate the mechanical ventilation treatment at the most appropriate time.

A significant portion of the extremely preterm babies may fail extubation even if the clinical criteria traditionally used for extubation are met. Unsuccessful extubation is associated with increased intraventricular bleeding, death, BPD, death or BPD, longer duration of ventilator support.

When respiratory failure and lung pathologies of extremely preterm babies begin to improve, the target for mechanical ventilation should be early and successful extubation. Currently, the decision to extubate a preterm baby is primarily based on clinical judgment. Only a few studies that showed the low predictive value and limited utility using different measures have evaluated readiness for extubation. Lung ultrasonography (USG) is a noninvasive bedside technique that has been found useful for predicting the success of weaning from the ventilator in adults; however, very little data are available in neonates. In a recently published study, it was proposed an extubation readiness estimation tool based on clinical and demographic data of preterm babies who were attempted elective extubation.

The researchers' hypothesis is that the use of a model based on extubation success scoring and lung USG scoring before extubation; reduces the failure of the first extubation attempt in very low birth weight infants. The aim of the study is to evaluate the value of using a model based on pre-extubation "extubation readiness predictor" and lung USG scoring to predict extubation success in preterm babies undergoing invasive mechanical ventilation.

This study is a prospective observational study. The study is planned to be conducted in infants with a birth weight <1250 g, who were intubated within the first 7 days of life, remained intubated invasive conventional mechanical ventilation for at least 48 hours, did not complete the postnatal 60 days, and met the traditional extubation criteria of the institution and were considered for elective extubation for the first time.

An "informed consent form" will be obtained from the parents of the babies included in the study. The birth dates, protocol numbers, birth types, maternal histories, genders, weeks of gestation and birth weights of the babies will be recorded.

The usual institutional routine approaches will be applied after the baby is born.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight <1250 gr
* Being intubated within the first 7 days of life and then followed on mechanical ventilation
* Being intubated for at least 48 hours
* Not completing the postnatal 60 days
* Meeting conventional clinical extubation criteria
* Having planned extubation for the first time
* Having no air leakage occurred
* Having no structural heart and lung disease
* Having no congenital and chromosomal anomalies
* Having an intact diaphragm
* Having no PVL, IVH (Grade 2 and above), HIE, meningitis or known CNS anomaly during extubation

Exclusion Criteria:

* Infants with a gestational age of 34 weeks or more
* Infants with unplanned and spontaneous extubation
* Infants who have tried extubation before
* Infants with hydrops fetalis
* Infants with chest deformities
* Infants with central respiratory failure (insufficient respiratory effort/control or continuous apneic)
* Infants who are neurologically depressed and do not have spontaneous breathing (hypocarbia due to hyperventilation, presence of severe sedation, use of neuromuscular drugs)
* In the presence of genetic or congenital anomalies (esophageal atresia, severe diaphragmatic hernia, diaphragm paralysis)
* Having phrenic nerve damage
* Presence of congenital myopathy
* Having any air leakage
* Having structural heart and lung disease
* Having no intact diaphragm
* Having PVL, IVH (Grade 2 and above), HIE, meningitis or known CNS anomaly during extubation

Ages: 48 Hours to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All premature infants with planned extubation during the study period.
Sampling Method: Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-04-20 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Extubation success | For at least 5 days during the post-extubation period.
  Not to be reintubated for at least 5 days during the post-extubation period.

SECONDARY OUTCOMES:
The incidence of morbidities related with prematurity. | 40 weeks' postmenstrual age.
  The incidence of morbidities related with prematurity (e.g. bronchopulmonary dysplasia, death and/or BPD, air leak syndromes, necrotizing enterocolitis, grade II and higher Intraventricular hemorrhage, retinopathy of prematurity, patent ductus arteriosus).
  Bronchopulmonary dysplasia will be assessed by attending clinicians based on the diagnostic criteria 2001 NICHD.
  * Air leaks will be assessed by chest X-ray.
  * Necrotizing enterocolitis will be assessed by abdominal X-ray and abdominal ultrasonography.
  * Intraventricular hemorrhage will be assessed by cranial ultrasonography.
  * Retinopathy of prematurity will be assessed by an expert ophthalmologist.
  * Patent ductus arteriosus will be assessed by echocardiography which will be performed by a pediatric cardiologist.
Length of stay in the hospital. | 40 weeks' postmenstrual age.
  Length of stay in the hospital.
Time elapsed on mechanical ventilation among survivors and the time taken with supplemental oxygen. | 40 weeks' postmenstrual age.
  Time elapsed on mechanical ventilation among survivors and the time taken with supplemental oxygen.
Total noninvasive support time. | 40 weeks' postmenstrual age.
  Total noninvasive support time until 40 weeks' postmenstrual age.
Percentage of time spent below 90% and above 95% on the SpO2 histogram. | During the first 5 days of the post-extubation period.
  Percentage of time spent below 90% and above 95% on the SpO2 histogram during the first 5 days of the post-extubation period.
Time to re-intubation in babies who are reintubated after extubation. | During the first 5 days of the post-extubation period.
  Time to re-intubation in babies who are reintubated after extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Eren Ozek, Study Director — Marmara University
Locations (2):
- Turkey (Türkiye) (2):
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Basaksehir Cam and Sakura City Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shi Y, Muniraman H, Biniwale M, Ramanathan R. A Review on Non-invasive Respiratory Support for Management of Respiratory Distress in Extremely Preterm Infants. Front Pediatr. 2020 May 28;8:270. doi: 10.3389/fped.2020.00270. eCollection 2020. PMID 32548084
- [Background] El Amrousy D, Elgendy M, Eltomey M, Elmashad AE. Value of lung ultrasonography to predict weaning success in ventilated neonates. Pediatr Pulmonol. 2020 Sep;55(9):2452-2456. doi: 10.1002/ppul.24934. Epub 2020 Jul 8. PMID 32609928
- [Background] Brat R, Yousef N, Klifa R, Reynaud S, Shankar Aguilera S, De Luca D. Lung Ultrasonography Score to Evaluate Oxygenation and Surfactant Need in Neonates Treated With Continuous Positive Airway Pressure. JAMA Pediatr. 2015 Aug;169(8):e151797. doi: 10.1001/jamapediatrics.2015.1797. Epub 2015 Aug 3. PMID 26237465
- [Background] Gupta D, Greenberg RG, Sharma A, Natarajan G, Cotten M, Thomas R, Chawla S. A predictive model for extubation readiness in extremely preterm infants. J Perinatol. 2019 Dec;39(12):1663-1669. doi: 10.1038/s41372-019-0475-x. Epub 2019 Aug 27. PMID 31455825